CLINICAL TRIAL: NCT01395927
Title: An Open-Label, Fixed-Sequence Study to Assess Effects of Steady-State Rifampin on the Single-Dose Pharmacokinetics of Canagliflozin in Healthy Subjects
Brief Title: A Study to Evaluate the Effects of Rifampin on Single-Dose Pharmacokinetics of Canagliflozin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CR018604; 28431754DIA1029
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
Keywords: Canagliflozin; Rifampin; Pharmacokinetics
MeSH Terms: interventions — Rifampin; Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): Canagliflozin Type=1 unit=mg number=300 form=tablet. Single dose of one 300-mg tablet on Day 1 and Day 10,Rifampin Type=2 unit=mg number=300 Form=capsule route=oral use. Two 300-mg capsules once daily on days Days 4 through 12.
  Interventions: Drug: Rifampin; Drug: Canagliflozin

INTERVENTIONS:
Drug: Rifampin — Type=2, unit=mg, number=300, Form=capsule, route=oral use. Two 300-mg capsules once daily on days Days 4 through 12.
Drug: Canagliflozin — Type=1, unit=mg, number=300, form=tablet. Single dose of one 300-mg tablet on Day 1 and Day 10

SUMMARY:
The purpose of this study is to evaluate blood levels of canagliflozin in healthy volunteers before and after the administration of multiple-doses of rifampin.

DETAILED DESCRIPTION:
This is an open-label (volunteer and study staff will know the identity of study drugs assigned) study of canagliflozin and rifampin taken in a sequential order by healthy volunteers for up to 12 days. Healthy volunteers will take orally (by mouth) one 300 mg canagliflozin tablet and/or two 300 mg rifampin capsules daily in sequential order as follows: on Day 1 volunteers will take one 300-mg canagliflozin tablet, on Days 4 to 9 volunteers will take two 300-mg rifampin capsules once daily, on Day 10 volunteers will take one 300-mg canagliflozin tablet + two 300-mg rifampin capsules, and on Days 11 and 12 volunteers will take two 300-mg rifamplin capsules once daily.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with a body mass index between 18 and 30 kg/m2 (inclusive)

Exclusion Criteria:

* History of or current medical illness deemed clinically significant by the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of canagliflozin | Day 1 up to Day 13

SECONDARY OUTCOMES:
Plasma concentrations of Rifampin | Day 9 up to Day 13
Adverse events reported | For approximately 13 days

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Overland Park, Kansas, United States